CLINICAL TRIAL: NCT03190629
Title: The Effect of On-line Hemodiafiltratrion on Nutritional Status and Body Composition: A Prospective, Controlled, Pilot Study
Brief Title: The Effect of On-line Hemodiafiltratrion on Nutritional Status and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pablo Molina (Other)
Responsible Party: Sponsor-Investigator, Pablo Molina, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OL-HDF-63/16
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: body composition; bioimpedance; hemodialysis; hemodiafiltration; nutritional status; protein energy wasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flux hemodialysis (Active Comparator): 3 times per week
  Interventions: Device: High-flux hemodialysis
- On line-hemodiafiltration (Experimental): 3 times per week
  Interventions: Device: On line-hemodiafiltration

INTERVENTIONS:
Device: High-flux hemodialysis — Hemodialysis treatment thrice weekly with the high-flux FX-100 dialyzer (Fresenius Medical Care, Bad Homburg, Germany; membrane: Helixone®; surface: 2.2 m2; UF coefficient: 73 ml/h mm Hg; ß2-microglobulin-sieving coefficient: 0.8; albumin-sieving coefficient: 0.001), including a minimum target dialysis dose (Kt/Vurea) ≥1.2 and a session length of 3.0 to 6.0 h. Hemodialysis treatments were performed with the 5008 hemodialysis system (Fresenius Medical Care).
  Arms: High-flux hemodialysis
Device: On line-hemodiafiltration — Post-dilution on line-hemodiafiltration treatment thrice weekly with the high-flux FX-100 dialyzer (Fresenius Medical Care, Bad Homburg, Germany; membrane: Helixone®; surface: 2.2 m2; UF coefficient: 73 ml/h mm Hg; ß2-microglobulin-sieving coefficient: 0.8; albumin-sieving coefficient: 0.001), including a minimum target dialysis dose (Kt/Vurea) ≥1.2 and a session length of 3.0 to 6.0 h. Post-dilution on line-hemodiafiltration treatments were performed with the 5008 hemodialysis system (Fresenius Medical Care), with automatic adjustment of the substitution fluid flow rate for maximising substitution volume while simultaneously avoiding haemoconcentration and filter clotting.
  Arms: On line-hemodiafiltration

SUMMARY:
Compared to conventional hemodialysis (HD), on-line hemodiafiltration (OL-HDF) achieves a more efficient removal of uremic toxins and reduces inflammation, which could favourably affect nutritional status. The aim of this study was to evaluate the 1-year effect of OL-HDF on nutritional status and body composition in prevalent HD patients.

DETAILED DESCRIPTION:
Postdilution on-line hemodiafiltration (OL-HDF) is considered the most efficient renal replacement treatment modality. Compared with conventional hemodialysis (HD), OL-HDF enables a better removal of middle molecular weight uremic toxins by combining convective and diffusive clearance. Although higher convection volume exchange has been associated with an increased survival advantage for dialysis patients, the mechanisms by which OL-HDF may improve outcomes remain unknown.

On the basis of improved toxin removal, a potential benefit of OL-HDF on nutritional status has been postulated. However, evidence on the effect of OL-HDF on nutritional status is scarce and at times conflicting. Some observational and interventional studies have suggested that OL-HDF is associated with improved nutritional parameters; others have found no effect; and one study even reported negative effects of OL-HDF on nutritional status. The majority of these observations come from cohort studies, non-controlled interventions and/or secondary analysis of controlled trials. Further, there are currently no data examining the plausible effect of postdilution OL-HDF on body composition. To clarify this important knowledge gap, this prospective, controlled, study evaluated the effects of high volume postdilution OL-HDF on nutritional status and body composition in prevalent HD patients.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 yr old; receiving stable high-flux hemodialysis treatment for at least 3 mo (Kt/Vurea ≥1.2 and hemodialysis performed 3.0 to 6.0 h, three times weekly), and agreed to give informed consent.

Exclusion Criteria:

* malabsorption syndrome; active malignant disease or other critical illnesses; or treated with steroids or antiandrogens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-03-31 (Actual)

PRIMARY OUTCOMES:
Lean tissue mass in kilograms | Baseline, 4, 8, and 12 months.
  Change from baseline to end of study in lean tissue mass in kilograms, measured quarterly throughout the 12-month intervention. Lean tissue mass was assessed by multi-frequency bioimpedance spectroscopy (Fresenius Medical Care) by experienced research staff blinded to all clinical and biochemical data of the patients. In order to control for potential variability and the effect of overhydration, all bioimpedance analyses were performed before a mid-week dialysis session.
Intracellular water in liters | Baseline, 4, 8, and 12 months.
  Change from baseline to end of study in intracellular water in liters, measured quarterly throughout the 12-month intervention. Intracellular water was assessed by multi-frequency bioimpedance spectroscopy (Fresenius Medical Care) by experienced research staff blinded to all clinical and biochemical data of the patients. In order to control for potential variability and the effect of overhydration, all bioimpedance analyses were performed before a mid-week dialysis session.
Body cell mass in kilograms | Baseline, 4, 8, and 12 months.
  Change from baseline to end of study in body cell mass in kilograms, measured quarterly throughout the 12-month intervention. Body cell mass was assessed by multi-frequency bioimpedance spectroscopy (Fresenius Medical Care) by experienced research staff blinded to all clinical and biochemical data of the patients. In order to control for potential variability and the effect of overhydration, all bioimpedance analyses were performed before a mid-week dialysis session.

SECONDARY OUTCOMES:
Serum prealbumin levels in milligrams per deciliter | Baseline, 4, 8, and 12 months.
  Change from baseline to end of study in serum prealbumin concentration in milligrams per decilitre, measured quarterly throughout the 12-month intervention. Pre-dialytic blood samples were collected after insertion of the access needle, and the post-dialytic sample was drawn from the arterial needle after slowing the blood punt to 50 ml/min. Prealbumin was determined by nephelometry with the IMMAGE800 Immunochemistry System (Beckman Coulter, Galway, Ireland).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Molina, MD, PhD, Principal Investigator — Department of Nephrology, Hospital Universitari Dr Peset, Department of Medicine, Universitat de València, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gatti E, Ronco C. Seeking an optimal renal replacement therapy for the chronic kidney disease epidemic: the case for on-line hemodiafiltration. Contrib Nephrol. 2011;175:170-185. doi: 10.1159/000333636. Epub 2011 Dec 15. PMID 22188699
- [Background] Canaud B, Bowry SK. Emerging clinical evidence on online hemodiafiltration: does volume of ultrafiltration matter? Blood Purif. 2013;35(1-3):55-62. doi: 10.1159/000345175. Epub 2013 Jan 22. PMID 23343547
- [Background] Fischbach M, Terzic J, Menouer S, Dheu C, Seuge L, Zalosczic A. Daily on line haemodiafiltration promotes catch-up growth in children on chronic dialysis. Nephrol Dial Transplant. 2010 Mar;25(3):867-73. doi: 10.1093/ndt/gfp565. Epub 2009 Nov 4. PMID 19889872
- [Background] Maduell F, Navarro V, Rius A, Torregrosa E, Sanchez JJ, Saborit ML, Ferrero JA. [Improvement of nutritional status in patients with short daily on-line hemodiafiltration]. Nefrologia. 2004;24(1):60-6. Spanish. PMID 15083959
- [Derived] Molina P, Vizcaino B, Molina MD, Beltran S, Gonzalez-Moya M, Mora A, Castro-Alonso C, Kanter J, Avila AI, Gorriz JL, Estan N, Pallardo LM, Fouque D, Carrero JJ. The effect of high-volume online haemodiafiltration on nutritional status and body composition: the ProtEin Stores prEservaTion (PESET) study. Nephrol Dial Transplant. 2018 Jul 1;33(7):1223-1235. doi: 10.1093/ndt/gfx342. PMID 29370428